CLINICAL TRIAL: NCT01568047
Title: Multicentre, Double-blind, Randomised, Placebo-controlled Study in Four Parallel Groups of PD Patients Treated With Standard-release Levodopa/Carbidopa 100/25 mg (Sinemet®) or Levodopa/Benserazide 100/25 mg (Madopar®/Restex®) and With Motor Fluctuations ("Wearing-off" Phenomenon)
Brief Title: Multicentre Study in Four Parallel Groups of Parkinson's Disease (PD) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BIA-91067-202; 2009-012897-12 (EudraCT Number)
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Results first posted 2015-01-08 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-11

CONDITIONS: Parkinson's Disease
Keywords: Parkinson Disease; BIA 9-1067
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone; carbidopa, levodopa drug combination; Levodopa

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): PLC, Placebo
  Levodopa/Carbidopa combination were given to half of the volunteers and Levodopa/Benzerazide to the other half
  Interventions: Drug: Placebo; Drug: Levodopa/Carbidopa; Drug: Levodopa/Benzerazide
- BIA 9-1067 - 5 mg (Experimental): 5 mg BIA 9-1067 (OPC, Opicapone)
  Levodopa/Carbidopa combination were given to half of the volunteers and Levodopa/Benzerazide to the other half
  Interventions: Drug: BIA 9-1067; Drug: Levodopa/Carbidopa; Drug: Levodopa/Benzerazide
- BIA 9-1067 - 15 mg (Experimental): 15 mg BIA 9-1067 (OPC, Opicapone)
  Levodopa/Carbidopa combination were given to half of the volunteers and Levodopa/Benzerazide to the other half
  Interventions: Drug: BIA 9-1067; Drug: Levodopa/Carbidopa; Drug: Levodopa/Benzerazide
- BIA 9-1067 - 30 mg (Experimental): 30 mg BIA 9-1067 (OPC, Opicapone)
  Levodopa/Carbidopa combination were given to half of the volunteers and Levodopa/Benzerazide to the other half
  Interventions: Drug: BIA 9-1067; Drug: Levodopa/Carbidopa; Drug: Levodopa/Benzerazide

INTERVENTIONS:
Drug: Placebo — once-daily
  Other Names: PLC
  Arms: Placebo
Drug: BIA 9-1067 — BIA 9-1067 - 5 mg single-dose
  Other Names: OPC, Opicapone
  Arms: BIA 9-1067 - 5 mg
Drug: BIA 9-1067 — BIA 9-1067 - 15 mg single-dose
  Other Names: OPC, Opicapone
  Arms: BIA 9-1067 - 15 mg
Drug: BIA 9-1067 — BIA 9-1067 - 30 mg single-dose
  Other Names: OPC, Opicapone
  Arms: BIA 9-1067 - 30 mg
Drug: Levodopa/Carbidopa — Levodopa 100 mg Carbidopa 25 mg
  Other Names: Sinemet
Drug: Levodopa/Benzerazide — Levodopa 100 mg Benzerazide 25 mg
  Other Names: Madopar®/Restex®

SUMMARY:
The purpose of this study is to investigate the tolerability and the effect of BIA 9-1067 at steady-state on the levodopa pharmacokinetics in Parkinson's Disease (PD) patients treated with levodopa/dopa-decarboxylase inhibitor.

DETAILED DESCRIPTION:
Multicentre, double-blind, randomised, placebo-controlled study in four parallel groups of PD patients treated with standard-release levodopa/carbidopa 100/25 mg (Sinemet®) or levodopa/benserazide 100/25 mg (Madopar®/Restex®) and with motor fluctuations ("wearing-off" phenomenon)

ELIGIBILITY:
Inclusion Criteria:

At screening (admission to the baseline period):

* Male or female of non-childbearing potential (by reason of surgery or postmenopausal);
* Age ≥ 30 years;
* A diagnosis of PD according to the UK PDS Brain Bank diagnostic criteria (bradykinesia and at least one of the following: muscular rigidity, rest tremor and postural instability);
* Predictable signs of end-of-dose deterioration despite "optimal" levodopa/carbidopa or levodopa/benserazide therapy;
* Modified Hoehn and Yahr stage of less than 5 in the "off" state; mean duration of "off" state ≥ 1.5 h during waking hours (based on historical information);
* Results of clinical laboratory tests acceptable by the investigator (not clinically significant for the well-being of the patient or for the purpose of the study);
* Able and willing to give written informed consent.

At randomisation (completion of the baseline period):

* Been treated with a stable regimen of 3 to 8 doses per day of standard-release levodopa/carbidopa 100/25 mg (Sinemet®) or levodopa/benserazide 100/25 mg (Madopar®/Restex®) for at least 1 week prior to randomisation;
* Mean duration of "off" state ≥ 1.5 h during waking hours (average of recordings of last 3 evaluable days on patient's diary);
* Concomitant anti-Parkinsonian medication (other than apomorphine, entacapone or tolcapone) in stable doses for at least 4 weeks prior to admission.

Exclusion Criteria:

At screening (admission to the baseline period):

* Non-idiopathic parkinsonism (atypical parkinsonism, symptomatic parkinsonism, Parkinson-plus syndrome);
* Treated with entacapone, tolcapone, neuroleptics, antidepressants (except serotonin-specific reuptake inhibitors or imipramines [desipramine, imipramine, clomipramine and amitriptyline]), monoamine oxidase inhibitors (except selegiline up to 10 mg/day in oral formulation or 1.25 mg/day in buccal absorption formulation or rasagiline up to 1 mg/day) or antiemetics (except domperidone) within 2 weeks prior to admission;
* Treated with any investigational product within 1 month prior to admission (or within 5 half-lives, whichever is longer);
* A psychiatric or any medical condition that might place him/her at increased risk or interfere with assessments;
* Known hypersensitivity to any of the ingredients of the investigational products;
* A history of abuse of alcohol, drugs or medications within the last 2 years;
* A clinically relevant ECG abnormality;
* A history or current evidence of heart disease, including but not limited to myocardial infarction, angina, congestive heart failure and cardiac arrhythmia;
* Unstable concomitant disease being treated with changing doses of medication;
* A history or current evidence of any relevant disease in the context of this study, i.e., with respect to the safety of the patient (e.g., hepatic impairment) or related to the study conditions;
* A test positive for the HIV-1 or HIV-2 antibodies, or hepatitis B surface antigen (HbsAg), or hepatitis C antibody (HCVAb);
* Donated blood or received blood or blood products within the 6 months prior to admission;
* Pregnant, breast-feeding or of childbearing potential;
* Other condition or circumstance that, in the opinion of the investigator, may compromise the patient's ability to comply with the study protocol.

At randomisation (completion of the baseline period):

* Treated with levodopa/DDCI in a 10:1 ratio or in a controlled-release formulation during the baseline period;
* Treated with apomorphine during the baseline period;
* A clinically relevant ECG abnormality.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- Romania (3):
  - Department of Neurology C.M.D.T.A. NEOMED, Brasov
  - Department of Neurology-Quantum Medical Center, Bucharest
  - Clinica de Medicina Fizica si Recuperare Medicala-Spitalul Clinic Judetean de Urgenta Craiova, Craiova
- Ukraine (4):
  - Ukrainian State Scientific Research Institute of Medical and Social Problems of Disability, Department of Neurology and Adjustment Conditions, Dnipropetrovsk
  - Department No. 23 of Communal setting of medical care Kharkiv's regional clinical psychiatric hospital No. 3,, Kharkiv
  - Department of Neuroinfections and multiple sclerosis, SI "Institute of Neurology, Psychiatry and Narcology of AMS of Ukraine, Kharkiv
  - Department of Clinical Physiology and Pathology of Extrapyramidal Nervous System SI "Institute of Gerontology, AMS Ukraine", Kyiv

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: PLC, Placebo
- BIA 9-1067 (5 mg); BIA 9-1067 (15 mg); BIA 9-1067 (30 mg): OPC, Opicapone
Period: Overall Study
Arm/Group | Placebo | BIA 9-1067 (5 mg) | BIA 9-1067 (15 mg) | BIA 9-1067 (30 mg)
Started | 10 | 10 | 10 | 10
Completed | 9 | 9 | 9 | 9
Not Completed | 1 | 1 | 1 | 1
Not completed — Ineligibility | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- BIA 9-1067 (5 mg): 5 mg BIA 9-1067 - OPC, Opicapone
- BIA 9-1067 (15 mg): 15 mg BIA 9-1067 - OPC, Opicapone
- BIA 9-1067 (30 mg): 30 mg BIA 9-1067 - OPC, Opicapone
- Total: Total of all reporting groups
Arm/Group | Placebo | BIA 9-1067 (5 mg) | BIA 9-1067 (15 mg) | BIA 9-1067 (30 mg) | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 40
Age, Customized [Number; unit: participants]
  ≤ 49 years | 0 | 0 | 0 | 0 | 0
  Between 49 and 88 years | 10 | 10 | 10 | 10 | 40
  ≥ 88 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 4 | 5 | 20
  Male | 5 | 4 | 6 | 5 | 20

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Observed Maximum Concentration
Description: Baseline period - to be switched respectively to standard-release levodopa/carbidopa 100/25 mg (Sinemet®) or levodopa/benserazide 100/25 mg (Madopar®/Restex®) and to adjust the number of daily doses.
  Test Period - After the baseline period during the 21 to 28 days
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- BIA 9-1067 5 mg: 5 mg BIA 9-1067 - OPC, Opicapone
- BIA 9-1067 15 mg: 15 mg BIA 9-1067 - OPC, Opicapone
- BIA 9-1067 30 mg: 30 mg BIA 9-1067 - OPC, Opicapone
Arm/Group | Placebo | BIA 9-1067 5 mg | BIA 9-1067 15 mg | BIA 9-1067 30 mg
Number analyzed (Participants) | 9 | 9 | 9 | 9
ng/mL
  Cmax (levodopa) Baseline | 1484 (26.0) | 1446 (37.6) | 1753 (43.4) | 1832 (49.1)
  Cmax (levodopa) Test | 1203 (29.4) | 1868 (31.8) | 1806 (28.4) | 2584 (33.7)
  Cmax (3-OMD) Baseline | 4701 (46.7) | 4631 (31.6) | 3529 (50.7) | 6222 (63.6)
  Cmax (3-OMD) Test | 3770 (45.0) | 2633 (21.2) | 1197 (71.8) | 1603 (36.2)
  Cmax (BIA 9-067) Test | NA (NA) — BIA 9-067 was not administered | 240 (186) | 233 (71.8) | 480 (64.4)

2. Secondary Outcome: AUC0-6 - Area Under the Plasma Concentration-time Curve (AUC) From Time Zero to to 6 h Postdose (AUC [0-6])
Description: as for outcome 1
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Placebo | BIA 9-1067 5 mg | BIA 9-1067 15 mg | BIA 9-1067 30 mg
Number analyzed (Participants) | 9 | 9 | 9 | 9
ng.h/mL
  AUC0-6 (levodopa) Baseline | 2841 (30.6) | 3451 (45.2) | 2734 (50.4) | 3862 (35.1)
  AUC0-6 (levodopa) Test | 2510 (27.7) | 4041 (18.3) | 4044 (38.7) | 6297 (25.5)
  AUC0-6 (3-OMD) Baseline | 23301 (39.7) | 23934 (28.3) | 18748 (58.8) | 34177 (61.9)
  AUC0-6 (3-OMD) Test | 21228 (45.4) | 14883 (22.2) | 6685 (73.1) | 9059 (36.5)
  AUC0-6 (BIA 9-067) Test | NA (NA) — BIA 9-067 was not administered | 627 (202) | 698 (73.1) | 1188 (54.8)

3. Primary Outcome: Tmax - Time to Observed Maximum Concentration
Description: as for outcome 1
Time Frame: 28 days
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Placebo | BIA 9-1067 5 mg | BIA 9-1067 15 mg | BIA 9-1067 30 mg
Number analyzed (Participants) | 9 | 9 | 9 | 9
ng/mL
  Cmax (levodopa) Baseline | 1.0 [0.5 to 4.0] | 1.0 [0.5 to 4.0] | 0.5 [0.5 to 1.0] | 1.0 [0.5 to 2.0]
  Cmax (levodopa) Test | 1.0 [0.5 to 2.0] | 1.0 [0.5 to 2.0] | 0.75 [0.5 to 2.0] | 0.5 [0.5 to 3.0]
  Cmax (3-OMD) Baseline | 2.0 [0.0 to 4.0] | 3.0 [1.0 to 6.0] | 2.25 [0.0 to 3.0] | 3.0 [0.0 to 6.0]
  Cmax (3-OMD) Test | 2.0 [0.0 to 6.0] | 1.5 [0.0 to 3.0] | 3.0 [2.0 to 4.0] | 3.0 [1.0 to 4.0]
  Cmax (BIA 9-067) Test | NA [NA to NA] — BIA 9-067 was not administered | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 4.0]

ADVERSE EVENTS:
Time Frame: 16 months
Groups:
- Placebo: Placebo, PLC
- BIA 9-1067 (5 mg): 5 mg BIA 9-1067, OPC, Opicapone
- BIA 9-1067 (15 mg): 15 mg BIA 9-1067, OPC, Opicapone
- BIA 9-1067 (30 mg): 30 mg BIA 9-1067, OPC, Opicapone
Arm/Group | Placebo | BIA 9-1067 (5 mg) | BIA 9-1067 (15 mg) | BIA 9-1067 (30 mg)
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 5/10 | 1/10 | 1/10 | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | BIA 9-1067 (5 mg) (N=10) | BIA 9-1067 (15 mg) (N=10) | BIA 9-1067 (30 mg) (N=10)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 1 | 1
TOOTHACHE (Gastrointestinal disorders) | 0 | 0 | 0 | 1
DRUG EFFECT DECREASED (General disorders) | 0 | 0 | 1 | 0
FATIGUE (General disorders) | 0 | 1 | 1 | 0
BLOOD CREATINE (Investigations) | 1 | 0 | 0 | 0
PHOSPHOKINASE INCREASED BLOOD LACTATE (Investigations) | 1 | 0 | 0 | 0
DEHYDROGENASE INCREASED BLOOD PRESSURE INCREASED (Investigations) | 1 | 0 | 0 | 0
DIZZINESS (Nervous system disorders) | 1 | 1 | 1 | 0
DYSKINESIA (Nervous system disorders) | 0 | 0 | 0 | 1
PARKINSON'S DISEASE (Nervous system disorders) | 0 | 0 | 1 | 0
TREMOR (Nervous system disorders) | 0 | 1 | 0 | 0
BRADYPHRENIA (Psychiatric disorders) | 0 | 0 | 1 | 0
DEPRESSION (Psychiatric disorders) | 0 | 0 | 1 | 0
INSOMNIA (Psychiatric disorders) | 1 | 0 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
SEBORRHOEIC DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
HYPERTENSION (Vascular disorders) | 1 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other